CLINICAL TRIAL: NCT06077981
Title: Comparison of 0.4% Hyaluronic Acid Solution Versus Hydroxyethylamide Solution in Submucosal Endoscopic Resections of Superficial Malignant Esophageal Neoplasms: a Randomized Clinical Trial.
Brief Title: Comparison of 0.4% Hyaluronic Acid Solution Versus Hydroxyethylamide Solution in Submucosal Endoscopic Resections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Fauze Maluf Filho, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NP3042/22
Record Dates: First submitted 2023-09-27; First posted 2023-10-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Neoplasms; Endoscopic Mucosal Resection; Hyaluronic Acid
Keywords: Esophageal Neoplasms; Endoscopic Mucosal Resection; Hyaluronic Acid
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Randomization shall consist of 30 patients, of which:
  15 will be from the hydroxyethylamide Group, where the submucosal endoscopic dissection will be performed with submucosal injection of hydroxyethylamide.
  15 will be from the Hyaluronic acid group (TS-905 Blue Eye), where the submucosal endoscopic dissection with submucosal injection of hyaluronic acid (TS-905 Blue Eye) will be performed.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxyethylamide Group (Active Comparator): 15 will be from the hydroxyethylamide Group, where the submucosal endoscopic dissection will be performed with submucosal injection of hydroxyethylamide.
  Interventions: Procedure: Submucous Endoscopic Dissection with hydroxyethylamide
- Hyaluronic acid group (TS-905 Blue Eye) (Active Comparator): 15 will be from the Hyaluronic acid group (TS-905 Blue Eye), where the submucosal endoscopic dissection with submucosal injection of hyaluronic acid (TS-905 Blue Eye) will be performed.
  Interventions: Procedure: Submucous Endoscopic Dissection with Hyaluronic acid (TS-905 Blue Eye)

INTERVENTIONS:
Procedure: Submucous Endoscopic Dissection with hydroxyethylamide — The resection will be performed in three stages using hydroxyethylamide : delimitation, incision and dissection. Initially we will inject the hydroxyethylamide and examine the delimitation of the lesion. With Knife itself, using soft or Forced coagulation current, we will circumvent the limits of the lesion with punctual coagulations 5 mm away from it.
  Arms: Hydroxyethylamide Group
Procedure: Submucous Endoscopic Dissection with Hyaluronic acid (TS-905 Blue Eye) — The resection will be performed in three stages using Hyaluronic acid (TS-905 Blue Eye) : delimitation, incision and dissection. Initially we will inject the Blue-Eyed and examine the delimitation of the lesion. With Knife itself, using soft or Forced coagulation current, we will circumvent the limits of the lesion with punctual coagulations 5 mm away from it.
  Arms: Hyaluronic acid group (TS-905 Blue Eye)

SUMMARY:
This is a randomized, single-center clinical trial that will compare the efficacy of two substances used in the submucosal cushion formation stage of endoscopic submucosal resections of early esophageal malignant neoplasms. Such substances are hyaluronic acid in the form of TS-905 Blue Eyeₒ and hydroxyethylamide (Voluven®).

DETAILED DESCRIPTION:
1. Design of the study:

   This is a randomized clinical trial in a single center. The lesions will be randomized into three blocks based on the diameter of the largest axis (less than 3 cm, between 3 - 5 cm and greater than 5 cm).
2. Selection of patients:

   The population studied will be patients with early esophageal neoplasia diagnosed and/or referred for submucosal endoscopic dissection at the São Paulo Cancer Institute (ICESP), University of São Paulo.
3. Evaluation of effectiveness and definitions:

Effectiveness will be measured from the degree of usefulness. The degree of utility will be determined from two variables: obtaining or not a complete block resection and additional number of submucosal injections performed during endoscopic dissection. The solution that results in a complete block resection with a number of additional injections of 0 (excellent utility degree) or 1 (good utility degree) will be considered effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Superficial esophageal adenocarcinoma or squamous cell carcinoma with indication of ESD after discussion in a multidisciplinary oncological board
* Signed informed consent form

Exclusion Criteria:

* Residual or recurrent esophageal lesions
* Ulcerated esophageal lesions
* Patients with severe cardiovascular, kidney or liver disease
* History of hypersensitivity to hyaluronic acid
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Volume of solution | During the procedure
  Compare the volume of TS-905 Blue Eye versus the solution of hydroxyethylamide used.

SECONDARY OUTCOMES:
Procedure duration in minutes | During the procedure
  Evaluate how the procure lasts using each one of the solutions
Number of additional injections | During the procedure
  Evaluate the number of additional injections need to complete the lesion ressection

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo, Brazil